CLINICAL TRIAL: NCT02084459
Title: The Use of Guided Self-determination in the Treatment of Chronic Pain Patients Will Increase Life Skills and Thereby Life Quality of the Chronic Pain Patient
Brief Title: Guided Self-determination in the Treatment of Chronic Pain to Promote the Life Skills of the Patient
Acronym: GSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Collaborators: Naestved Hospital (Other); Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Anne Pickering, Nurse, project leader, Herlev Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HEH201300702085
Record Dates: First submitted 2014-03-03; First posted 2014-03-12 (Estimated); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Chronic Pain
Keywords: Chronic pain; Supportive care; Psychosocial Circumstances; Autonomy support; Nursing intervention
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Standard of care
- Autonomy-supportive counselling (GSD) (Experimental): GSD, an educational method, comprising 32 semi-structured reflection sheets inviting the patients in groups of 4 through 8 sessions of 150 minutes' duration to reflect on the patient's own situation and to be active in co-operation with the nurses.
  Interventions: Behavioral: Autonomy-supportive counselling (GSD)

INTERVENTIONS:
Behavioral: Autonomy-supportive counselling (GSD) — GSD, an educational method, comprising 32 semi-structured reflection sheets inviting the patients in groups of 4 through 8 sessions of 150 minutes' duration to reflect on the patient's own situation and to be active in co-operation with the nurses.
  Arms: Autonomy-supportive counselling (GSD)

SUMMARY:
The purpose of this randomized study is to find out whether using the Danish-developed nursing intervention guided self-determination (GSD) can improve life skills of the chronic pain patient.

The hypothesis is "using guided self-determination in the treatment of chronic pain patients will increase the life skills of the patients and thus their life quality in spite of pain".

DETAILED DESCRIPTION:
Twenty percent of the Danish population suffer from chronic pain, which leads to the second highest financial expense following psychiatric diseases. In treating chronic pain, the main focus is often on diagnosis and treatment rather than life quality and everyday life. Several studies point to the fact that the interaction between the health professional and the patient can be improved by the individual patient being educated in taking responsibility for his/her own illness, and by involving the patient in decision making through training communication.

GSD is an educational method, comprising 32 semi-structured reflection sheets inviting the patients in groups of 4 through 8 sessions of 150 minutes' duration to reflect on the patient's own situation and to be active in co-operation with the nurses.

A total of 192 patients will be included and randomized in either an intervention or in a control group. The difference between the two groups is measured by means of three questionnaires, SF-36, PAM and SOC, which are answered before and after the intervention as well as 6 months later.

The hypothesis is "using guided self-determination in the treatment of chronic pain patients will increase the life skills of the patients and thus their life quality in spite of pain".

An alliance is established between The Multidisciplinary Pain Clinic at Herlev Hospital and The Pain Clinic at Naestved Hospital as well as The Regional Pain Clinic at Koege Hospital to conduct this intervention and thus make the best possible use of interrelated knowledge within the issue.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older, diagnosed with nonmalignant chronic pain

Exclusion Criteria:

* patients who do not read, write and understand the Danish language
* patients with a known medical abuse
* patients needing special psychological and/or psychiatric intervention
* patients with health-related problems preventing them from participating in a group

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-02; Primary Completion 2016-07-15 (Actual); Study Completion 2016-07-15 (Actual)

PRIMARY OUTCOMES:
Changes in self-reported life quality | Baseline, 2, 6 months
  Measured by the self-rating "SF-36 (Short-form 36)" - questionnaire

SECONDARY OUTCOMES:
Changes in self-assessed motivation for pain management | Baseline, 2, 6 months
  Measured by the self-rating "PAM (Patient Activation Measure)"-questionnaire
Changes in self-assessed competence in pain management | Baseline, 2, 6 months
  Measured by the self-rating "SOC (Sense of Coherence)" - questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Mette Husum, RN, Principal Investigator — Herlev Hospital; Niels-Henrik Jensen, MD, Study Chair — Herlev Hospital
Locations (1):
- Herlev Hospital, Herlev, Danmark, Denmark

REFERENCES:
- [Derived] Pickering AP, Bache NJ, Estrup S. Guided self-determination in treatment of chronic pain - a randomized, controlled trial. Scand J Pain. 2021 Jul 31;22(2):288-297. doi: 10.1515/sjpain-2021-0007. Print 2022 Apr 26. PMID 34333889